CLINICAL TRIAL: NCT04335409
Title: Pneumonitis After Radiotherapy for Lung Cancer: A Symptom-Based Scoring System to Identify Patients Developing Radiation Pneumonitis
Brief Title: Pneumonitis After Radiotherapy for Lung Cancer
Acronym: PARALUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Prof Dirk Rades, Professor and Chair, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PARALUC
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pain Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants irradiated for lung cancer (Experimental): Participants who receive radiotherapy for lung cancer and have risk factors for developing radiation pneumonitis. Risk factors include mean dose to the ipsilateral lung >13 Gy plus at least one other factor (significant cardiovascular disease, history of heavy smoking (≥40 pack years), previous/concurrent chemotherapy or previous/adjuvant immunotherapy) or mean dose to the ipsilateral lung >20 Gy without other factors.
  Interventions: Diagnostic Test: Questionnaire; Other: Mobile Application

INTERVENTIONS:
Diagnostic Test: Questionnaire — The patients are asked to complete a questionnaire (paper version) once a week during the period of radiotherapy and up to 24 weeks following radiotherapy. In this questionnaire, the patients are asked to state and rate their symptoms potentially associated with pneumonitis. Scoring points are assigned to the severity of the symptoms (symptom scores), and the resulting sum score (patient score) will be used for identification of radiation pneumonitis.
Other: Mobile Application — In 10 patients, the paper version of the symptom-based scoring system (questionnaire) will be supplemented by a mobile application (app) asking the same questions regarding symptoms potentially associated with pneumonitis.

SUMMARY:
Major goals of radiotherapy include local disease control and improvement of the patients' prognoses. One possible side effect of radiotherapy for lung cancer is radiation pneumonitis. Severe (grade ≥3) radiation pneumonitis can even be fatal in approximately 2% of the patients. It would be important to identify patients developing radiation pneumonitis and requiring medical treatment early.

In the present study, the patients are asked to complete a questionnaire (paper version) once a week during the period of radiotherapy and up to 24 weeks following radiotherapy. In this questionnaire, the patients are asked to state and rate their symptoms potentially associated with pneumonitis. Scoring points are assigned to the severity of the symptoms (symptom scores), and the resulting sum score (patient score) will be used for identification of radiation pneumonitis.

The main goal of this trial is to evaluate the usefulness of a new symptom-based scoring system with respect to the identification of patients developing pneumonitis after radiotherapy of breast or lung cancer. The discriminative power of the symptom-based scoring system will be assessed by calculating the area under the ROC curve (AUC). Taking into account that 5% of patients will not qualify for Full Analysis Set, a total of 78 patients should be recruited.

If statistical significance of the AUC is reached, the most-informative (optimal) scoring point to identify radiation pneumonitis will be derived. Sensitivity analyses will be conducted to further investigate the performance of the symptom-based scoring system.

In 10 patients, the paper version of the symptom-based scoring system (questionnaire) will be supplemented by a mobile application (app) asking the same questions regarding symptoms potentially associated with radiation pneumonitis.

DETAILED DESCRIPTION:
Background Most patients with small-cell lung cancer (SCLC) receive radiotherapy in combination with chemotherapy as definitive treatment. Also, a considerable number of patients with advanced non-small-cell lung cancer (NSCLC) are treated with radiotherapy with or without concurrent chemotherapy. Radiation pneumonitis is a possible side effect of radiotherapy for lung cancer. Severe pneumonitis was reported to be fatal in approximately 2% of patients. In our centre, the prevalence of symptomatic radiation pneumonitis was 7.6% in patients irradiated for lung cancer. The prevalence of symptomatic radiation pneumonitis in patients with risk factors was 18.8%.

Pneumonitis can occur up to 23 weeks following radiotherapy. Therefore, the symptoms may not be associated with previous radiotherapy, and pneumonitis may be missed. It would be important to identify patients developing radiation pneumonitis and requiring medical treatment more early.

This study aims to develop a symptom-based scoring system that contributes to an earlier detection of radiation pneumonitis requiring medical intervention (grade ≥2) after radiotherapy for lung cancer. This scoring system is a prerequisite for a mobile application, which can be used by the patients at home to rate their symptoms possibly related to pneumonitis.

Patients are asked to complete a questionnaire (paper version) once a week during the period of radiotherapy and up to 24 weeks following radiotherapy. In this questionnaire, the patients are asked to state and rate their symptoms potentially associated with pneumonitis. Scoring points are assigned to the severity of the symptoms (symptom scores), and the resulting sum score (patient score) will be used for identification of radiation pneumonitis.

Primary endpoint To assess the performance characteristics of the symptom-based scoring system for detection of radiation pneumonitis the receiver operating characteristic (ROC) curve is used to show the connection between sensitivity and specificity for every possible cut-off for the scoring system and to select the optimal scoring point for detection of radiation pneumonitis- The area under the ROC curve (AUC) is calculated to prove the diagnostic ability of the scoring system.

General trial design and duration This is a single-center prospective study, which aims to assess the performance of a new symptom-based score and to identify its optimal scoring point with respect to the detection of patients developing pneumonitis following radiotherapy of breast cancer or lung cancer. The recruitment of all 98 patients (93 patients plus drop-outs) should be completed within 33 months. The treatment period will be 6-7 weeks, and the follow up period 24 weeks. This equals a total running time for the trial of approximately 40 months.

Symptom-Based Scoring System (Paper Version) The patients are asked to complete a paper-based questionnaire (symptom-based scoring system, paper version) once a week during the period of radiotherapy and up to 24 weeks following radiotherapy. The patients are asked to state and score their symptoms that are potentially associated with pneumonitis, namely cough, shortness of breath and fever. Scoring points are assigned to the severity of the symptoms (= symptom scores), and the resulting sum score (patient score) will be used to identify radiation pneumonitis.

During the time of radiotherapy, the patients will complete the paper-based questionnaire directly prior to their appointment with a physician who will perform a physical examination once a week. Following radiotherapy, the patients will be contacted by phone once a week and asked to answer the questions of the questionnaire.

In case of an increase of the total score compared to baseline, patients receive either a follow-up telephone call after 3 days, are asked to come to the hospital as outpatients or are admitted to hospital. In case of suspected pneumonitis, patients undergo lung function tests. If the suspected diagnosis of pneumonitis is substantiated, patients receive a chest x-ray plus/minus computed tomography. If the diagnosis symptomatic radiation pneumonitis (grade ≥2) has been confirmed, patients receive medical intervention. The vast majority of the patients receive prednisolone, which is considered the mainstay of the treatment for radiation pneumonitis.

The symptom-based sum score is correlated to pneumonitis (yes vs. no). At the end of radiotherapy, patients are asked to complete a questionnaire regarding their satisfaction with the score. In case of a dissatisfaction rate >20%, the score needs modifications before it can be used in future studies. In case of a dissatisfaction rate >40%, it will be considered not useful.

Subgroup Analysis: Symptom-Based Scoring System (Mobile Application) In 10 patients, the paper version of the symptom-based scoring system (questionnaire) will be supplemented by a mobile application (app) asking the same questions regarding cough, shortness of breath and fever. The symptoms collected by the app will not be evaluated or analyzed. With regard to the app, only its functionality will be tested in this study. The patients will be asked to complete the questionnaire of the app directly after completing the questionnaire of the paper version.

Statistics / Sample size calculation The main goal of this trial is to evaluate the usefulness of a new symptom-based scoring system with respect to the identification of patients developing pneumonitis after radiotherapy for lung cancer. The discriminative power of the symptom-based scoring system will be assessed by calculating the area under the ROC curve (AUC). Assuming a ratio between patients without and with radiation pneumonitis of 3.63, a sample size of 93 patients is required in the full analysis set to yield statistical significance at the significance level of 5% with a power of 90% if the AUC under the alternative hypothesis is in fact at least 0.9. Taking into account that 5% of patients will not qualify for Full Analysis Set, a total of 98 patients should be recruited.

If statistical significance of the AUC is reached, the most-informative (optimal) scoring point to identify radiation pneumonitis will be derived. Sensitivity analyses will be conducted to further investigate the performance of the symptom-based scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven lung cancer
2. Indication for radiotherapy
3. Risk factors for developing radiation pneumonitis
4. Age ≥18 years
5. Written informed consent
6. Capacity of the patient to contract

Exclusion Criteria:

1. Pregnancy, Lactation
2. Expected non-compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Grade ≥2 Radiation Pneumonitis | 24 weeks following radiotherapy
  Radiation pneumonitis will been assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, MD, Principal Investigator — Department of Radiation Oncology, University of Lübeck, Germany
Locations (1):
- Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Ratzeburger Allee 160, 23562 Lübeck, Germany, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Werner EM, Glatzel E, Eggert MC, Olbrich D, Tvilsted S, Bohnet S. Pneumonitis after radiotherapy for lung cancer (PARALUC): an interventional study to create a symptom-based scoring system for identification of patients developing radiation pneumonitis. BMC Cancer. 2020 Aug 20;20(1):785. doi: 10.1186/s12885-020-07291-5. PMID 32819311

DOCUMENTS (1):
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT04335409/ICF_000.pdf